CLINICAL TRIAL: NCT03023605
Title: Adherence to Clinical Guidelines in the Diagnosis of Pulmonary Embolism in an Emergency Department. Analysis of the Clinical Impact of a Training Intervention (APEED)
Brief Title: Analysis of a Training Intervention for Pulmonary Embolism Diagnosis in Emergency Department (APEED)
Acronym: APEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-EPU-2016-61
Record Dates: First submitted 2017-01-02; First posted 2017-01-18 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Adherence to practice guidelines; Age-adjusted D-dimer; Clinical prediction rules; Elderly patients
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention PE Diagnosis (No Intervention): Patients visited in Emergency Department, with suspected Pulmonary Embolism, before the training intervention.
- Post-intervention PE Diagnosis (Experimental): Patients visited in Emergency Department, with suspected Pulmonary Embolism, after the training intervention.
  Training intervention centered on emergency department staff, regarding the application of clinical probability scores (Wells and Geneva scores) to guide the determination of D-dimer and the performance of pulmonary CT in patients with suspected pulmonary embolism.
  Interventions: Behavioral: Training Intervention for PE Diagnosis

INTERVENTIONS:
Behavioral: Training Intervention for PE Diagnosis — Focused on the Emergency Department staff and the rotating residents during the months 4 and 5 of 2015, and consisted of:
  1. Clinical Update Sessions for staff ED (20 physicians)
  2. training sessions for residents that rotate in ED (60 physicians )
  3. Development of a triptych, including clinical prediction scales, combination algorithm of scales and D-Dimmer value
  4. Development of posters, with brief information
  5. Dissemination by e-mail of scientific information
  6. Direct reminder during the working day
  Arms: Post-intervention PE Diagnosis

SUMMARY:
The purpose of this study is to analyze the clinical impact of an educational intervention on adherence to Clinical Practice Guidelines in an Emergency Department (ED), by using a standardized training, for improving diagnostic sensibility and reducing unnecessary scans, adverse effects and stays in the ED.

DETAILED DESCRIPTION:
The Hospital de la Santa Creu i Sant Pau Emergency Department (ED) implemented a training program between May and June 2015 to improve compliance and adherence to recommended clinical practice and optimize the diagnosis and management of patients with suspected Pulmonary Embolism (PE). The training program was standardized, systematic and continuous, with subsequent reinforcement to ensure implementation. This paper aims to evaluate the clinical impact of the training intervention. The establishment of training measures to improve adherence to guidelines implies clinical practice improvement and benefits patients and health system. Moreover, it is a simple and inexpensive intervention, and can be easily reproduced in other ED.

All adult patients (<18 y) with suspected pulmonary embolism attended at Emergency Department will be included. Retrospective information from two different periods (before and after the training intervention) will be collected. First period: 1/1/2012 - 31/12/2012 and second Period: 01.06.2015 - 30/11/2015, pre and post intervention.

OBJECTIVES

A. Primary:

1. Analyze adherence to guidelines for the evaluation of suspected PE in the ED.
2. Determine the clinical impact of training intervention (change in adherence to guidelines after training measures among staff in Emergency Department)
3. Implementation and consolidation of a systematic, standardized, continuous training intervention for improving processes and results.

B.- Secondary

1. Analyze PE cases (presentation, clinical features, treatment, clinical evolution)
2. analyze the clinical differences in three subgroups of patients with PE: young patients (<50 years), elderly patients (<65 years) and cancer
3. Analyze the value of D-dimmer corrected by age in diagnostic algorithms
4. Analyze the results of a new algorithm (EPC + Dimmer corrected age) in the elderly population group (<65 years).

ELIGIBILITY:
Inclusion Criteria:

* Are included
* those patients who underwent a D-dimmer for suspected PE
* all those who underwent the diagnosis of PE at discharge
* those who died from EP.

Exclusion Criteria:

* Are excluded:
* all patients who underwent D-dimmer test with a different diagnosis of EP and those who had a chronic EP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of cases where clinical guidelines have been followed for suspected Pulmonary Embolism in the Emergency Department (adherence) | 3 months
  October, November, December 2016
Number of cases where clinical guidelines have been followed for suspected Pulmonary Embolism in the Emergency Department (adherence) after training measures among staff in Emergency Department | 3 months
  January, February and Mach 2017

SECONDARY OUTCOMES:
Prevalence of different clinical characteristics of Pulmonary Embolism (presentation, clinical features, treatment, clinical evolution) | 12 months
Prevalence of different clinical characteristics of Pulmonary Embolism related to age (three subgroups of patients with PE: young patients (<50 years), elderly patients (<65 years) and cancer) | 12 months
D-dimmer corrected by age in all cases | 12 months
Sensibility and Specificity of new algorithm (Clinical Score+ Dimmer corrected age) in the elderly population group (<65 years) | 12 months

OTHER OUTCOMES:
Adherence to clinical guidelines after the implementation of a systematic, standardized, continuous training intervention for improving processes and results. | 12 months
  Number of patients with suspected pulmonary embolism in whom the decision to perform D-Dimer and TC was based on clinical probability scores (Wells and Geneva test)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Puig, PhD, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau - IIB Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided